CLINICAL TRIAL: NCT06863363
Title: A Multicenter, Randomized, Open-label, Parallel-controlled Clinical Trial Comparing the Efficacy and Safety of PEG-rhGH Injection Combined with Semaglutide Injection Versus Semaglutide Injection Monotherapy in Body Composition of Non-Diabetic Obese Adults
Brief Title: PEG-rhGH and Semaglutide Combination Therapy in Non-Diabetic Obese Adults
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS24-B046-401
Record Dates: First submitted 2025-02-28; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Non-diabetic Obesity
MeSH Terms: interventions — polyethylene glycol-recombinant human growth hormone; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEG-rhGH Injection + Semaglutide Injection (Experimental)
  Interventions: Drug: PEG-rhGH Injection + Semaglutide Injection
- Semaglutide Injection (Active Comparator)
  Interventions: Drug: Semaglutide Injection

INTERVENTIONS:
Drug: PEG-rhGH Injection + Semaglutide Injection — Polyethylene Glycol Recombinant Human Growth Hormone Injection (PEG-rhGH Injection), 54 IU/9.0 mg/1.0 mL/amp.; Subcutaneous injection using pen-injector, once weekly at a dose of 2 mg per week (weeks 1-40).
  Semaglutide Injection, 0.68 mg/mL，1.5 mL；1.34 mg/mL，1.5 mL；1.34 mg/mL，3 mL；2.27 mg/mL，3 mL；3.2 mg/mL，3 mL; Subcutaneous injection once weekly using pre-filled pen including dosage escalation period (W1-W16): starting dose 0.25 mg, increasing every 4 weeks (0.25 mg, 0.5 mg, 1.0 mg, 1.7 mg, 2.4 mg) and maintenance treatment period (W17-W40): at a dose of 2.4 mg for 24 weeks
  Arms: PEG-rhGH Injection + Semaglutide Injection
Drug: Semaglutide Injection — Semaglutide Injection, 0.68 mg/mL，1.5 mL；1.34 mg/mL，1.5 mL；1.34 mg/mL，3 mL；2.27 mg/mL，3 mL；3.2 mg/mL，3 mL; Subcutaneous injection once weekly using pre-filled pen including dosage escalation period (W1-W16): starting dose 0.25 mg, increasing every 4 weeks (0.25 mg, 0.5 mg, 1.0 mg, 1.7 mg, 2.4 mg) and maintenance treatment period (W17-W40): at a dose of 2.4 mg for 24 weeks
  Arms: Semaglutide Injection

SUMMARY:
This study aims to evaluate the efficacy and safety of PEG-rhGH Injection combined with Semaglutide Injection versus Semaglutide Injection monotherapy in improving body composition (lean body mass, fat mass, etc.) in non-diabetic obese adults, while also analyzing changes in body weight, blood glucose, and other metabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 years (minimum age) and 50 years (maximum age), inclusive
2. Gender: Male or female, with a ratio of male to female being 2:1;
3. Body Mass Index (BMI) ≥28 kg/m²;
4. No prior use of semaglutide injection or antidiabetic medications;
5. Free Thyroxine (FT4) levels within normal range at screening;
6. Testosterone levels within normal range at screening (males only);
7. No plans for pregnancy from the time of signing the ICF until 2 months after the study ends, willingness to take effective contraceptive measures to prevent pregnancy or causing a partner's pregnancy, and no plans for sperm or egg donation during the study period;
8. Participants must voluntarily agree to and be able to comply with all scheduled visits, treatment plans, laboratory tests, special examinations, neurological assessments, and other trial procedures, and sign a written informed consent form.

Exclusion Criteria:

1. Unable to accept regular follow-up;
2. Those who have difficulty with self-injection;
3. Weight change >5.0% in the 12 weeks prior to screening (self-reported);
4. History of allergic reactions to the study drug or similar drugs;
5. Evaluated by the investigator as unable to tolerate subcutaneous injection, such as those undergoing anticoagulant therapy, thrombocytopenia, known bleeding disorders, or idiopathic thrombocytopenic purpura;
6. Planning surgery within 1 year; history of gastrointestinal surgery (excluding polypectomy and appendectomy);
7. Positive blood HCG during screening; breastfeeding women; postmenopausal women; women with FSH >30 IU/L during screening;
8. Any of the following: myocardial infarction, stroke, unstable angina requiring hospitalization, or transient ischemic attack within 180 days before screening, classified as NYHA class III or higher;
9. Clinically significant severe ECG abnormalities (e.g., QT prolongation [>450 ms in men, >470 ms in women], ventricular Flutter, ventricular fibrillation, torsades de pointes, sick sinus syndrome, third-degree heart block without pacemaker therapy, and other severe abnormalities as assessed by the investigator), uncontrolled blood pressure despite treatment/untreated (systolic BP ≥160 mmHg and/or diastolic BP ≥100 mmHg during screening, systolic BP <90 mmHg and/or diastolic BP <50 mmHg), or other cardiovascular diseases deemed unsuitable for the study by the investigator;
10. Triglycerides ≥500 mg/dL (5.65 mmol/L);
11. Current or past history of malignancy, or currently having nodules with malignant potential such as thyroid nodules with TIRADS grade ≥4;
12. Tumor markers during screening: CA125 (for women), CA199, CEA, AFP above upper limit of normal range; PSA above upper limit of normal range (for men);
13. Hemoglobin A1c ≥6.5% during screening;
14. History of diabetes (type 1, type 2, special types, or gestational diabetes) or currently using injectable or oral antidiabetic medications;
15. Current or past history of acromegaly;
16. Proliferative or severe non-proliferative diabetic retinopathy at screening; fundus examination within 90 days before randomization: proliferative retinopathy or macular edema requiring acute treatment;
17. Used growth hormone therapy in the past 6 months;
18. Used any weight loss medications in the past 3 months; previously underwent obesity surgery or planned obesity surgery during the study;
19. Any of the following laboratory tests at screening: AST or ALT >2.5 ULN; total bilirubin >1.5 ULN; TSH <0.4 or >6 mIU/L; calcitonin >50 ng/L;
20. IGF-1 SDS >2.0 (age and gender matched);
21. Serum creatinine >1.5 ULN, eGFR <60 mL/min/1.73 m² [using the modified simplified MDRD equation: eGFR = 175 × (serum creatinine in mg/dL)^-1.234 × age^-0.179 × 0.79 for women], or kidney impairment requiring dialysis;
22. History of pancreatitis, or current acute or chronic pancreatitis;
23. History of cholecystitis, or current gallbladder/biliary disease symptoms, or treatable gallstones or polyps;
24. Family or personal history of multiple endocrine neoplasia type 2 or thyroid cancer (family defined as first-degree relatives);
25. Prior history of pituitary mass;
26. History of seizures;
27. Participated in another clinical trial with approved or investigational drugs/devices within 90 days before screening (excluding those who only signed the consent without receiving any intervention);
28. History of substance abuse and/or alcoholism, or mental disorders; during screening, had impaired consciousness including somnolence, stupor, coma, confusion;
29. Questionnaire PHQ-9 score ≥15; history of suicidal behavior; Columbia-Suicide Severity Rating Scale (C-SSRS) question 1 or 2 indicating suicidal ideation (answering "yes" to question 1 or 2);
30. Other reasons for exclusion as deemed by the investigator, such as any situation endangering participant safety or affecting compliance with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 212 (Estimated)

PRIMARY OUTCOMES:
The change in lean body weight (kg) from baseline | Week 40

SECONDARY OUTCOMES:
Change in lean body mass percentage (%) | During 40 weeks
Change in appendicular muscle mass (kg) | During 40 weeks
Change in trunk muscle mass (kg) | During 40 weeks
Change in appendicular fat mass (kg) | During 40 weeks
Change in trunk fat mass (kg) | During 40 weeks
Percentage change in total fat mass (%) | During 40 weeks
Change in total fat mass (kg) | During 40 weeks
Waist circumference change (cm) | During 40 weeks
Body weight change (kg) | During 40 weeks
Glycated hemoglobin change (%) | During 40 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided